CLINICAL TRIAL: NCT05647018
Title: In-hospital Clinical Outcome of Deferred Stenting Versus Immediate Stenting in the Management of Acute STEMI Presenting With High Thrombus Burden: A Randomized Control Study
Brief Title: In-hospital Clinical Outcome of Deferred Stenting Versus Immediate Stenting in the Management of Acute STEMI Presenting With High Thrombus Burden.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yomna Mahmoud Shokry Abdelrehim, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPCI in STEMI
Record Dates: First submitted 2022-11-19; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Coronary Thrombosis
MeSH Terms: conditions — Coronary Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deferred stenting in STEMI patients with high thrombus burden undergoing primary PCI (Active Comparator)
  Interventions: Procedure: Primary Percutaneous coronary angiography
- Non-deferred stenting in STEMI patients with high thrombus burden undergoing primary PCI (Active Comparator)
  Interventions: Procedure: Primary Percutaneous coronary angiography

INTERVENTIONS:
Procedure: Primary Percutaneous coronary angiography — Percutaneous coronary intervention (PCI) refers to a family of minimally invasive procedures used to open clogged coronary arteries in patients presenting with myocardial infarction, through which installment of stents or intracoronary injection of drugs can take place.
  Other Names: Minimally invasive mechanical intervention

SUMMARY:
To compare the in hospital clinical outcomes in terms of efficacy and safety of deferred stenting versus non-deferred stenting in STEMI patients with high thrombus burden undergoing primary percutaneous intervention.

DETAILED DESCRIPTION:
Angiographically, intracoronary thrombus is defined as the presence of a filling defect with reduced contrast density or haziness. Angiographic evidence of thrombus can be seen in 91.6% of patients who present with STEMI(1). Large intracoronary thrombus has an incidence of 16.4% of patients with acute coronary syndrome (ACS).

Thrombus encountered in the setting of ACS has been correlated with acute complications during percutaneous coronary interventions including: 3 times higher MACE - ischemic complications, lower procedural success, higher distal embolization leading to slow/no flow, high mortality, ST elevation and longer hospital stays.

High thrombus burden can be defined using Yip's criteria:

1. Large infarct-related artery (visually estimated reference vessel diameter ≥ 4 mm)
2. Angiographic thrombus with the greatest linear dimension > 3 times the reference vessel diameter;
3. "Cutoff pattern" (lesion morphology with an abrupt cutoff without taper before the occlusion);
4. Accumulated thrombus (> 5 mm of linear dimension) proximal to the occlusion;
5. Floating thrombus proximal to the occlusion;
6. Persistent dye stasis distal to the obstruction. IF more than two criteria indicate the presence of very high thrombus burden.

PCI Strategies introduced in HIGH thrombus BURDEN include incorporation of both pharmacological and mechanical thrombus removal.

Immediate stenting of the culprit coronary artery may lead to high chances of the slow-flow/no-reflow phenomenon that leads to periprocedural MI and adverse cardiovascular events. Current studies show that routine deferred stenting has not been found beneficial except when careful patient selection is done where deferral may reduce the final infarct size.

Glycoprotein IIa/IIIb inhibitors have been used in such cases. Current guidelines recommend GPIIa/IIb as bailout therapy following PCI when massive thrombus is found: Class IIa. (6) The rationale in using intracoronary GPIIa/IIIb is that it can be more effective, faster and safer in terms of bleeding.

Deferred stenting is a method of dealing with thigh thrombus burden in STEMI patients. This means to wait 24-48 hour and delay stenting. During this time gap, patient receives intravenous tirofiban. This may be beneficial as the thrombus burden will reduce, minimizing the occurrence of the slow-flow/no-reflow phenomenon.

During coronary angiography the epicardial perfusion can be demonstrated using the TIMI grade flow where:

* TIMI 0 flow (no perfusion) complete blockage - absence of any antegrade flow (forward flow) beyond a coronary occlusion.
* TIMI 1 flow (penetration without perfusion) is faint antegrade coronary flow beyond the occlusion, with incomplete filling of the distal coronary bed.
* TIMI 2 flow (partial reperfusion) is delayed or sluggish antegrade flow with complete filling of the distal territory.
* TIMI 3 is normal flow which fills the distal coronary bed completely. (7) During Primary PCI, If TIMI 0-1 flow is encountered a technique called minimally invasive mechanical intervention (MIMI) can be employed to restore flow. This MIMI entails the use of a guidewire, an undersized balloon or thrombus aspiration to establish distal coronary flow.

ELIGIBILITY:
Inclusion Criteria:

1. TIMI 2-3 flow in the infarct related artery (IRA) with high thrombus burden at initial angiography.
2. TIMI 2-3 in the IRA with high thrombus burden after MIMI.

Exclusion Criteria:

1. TIMI 0-1 flow in the IRA after MIMI.
2. TIMI 2-3 in the IRA with low thrombus burden.
3. Contraindication or hypersensitivity to Tirofiban
4. High bleeding risk calculated using the CRUSADE score >50.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the method used in terms of TIMI flow | During in hospital stay up to 36 hours
  By TIMI III flow finding
Effectiveness of the method used in regards to ECG. | During in hospital stay up to 36 hours
  ECG: ST segment resolution immediately after PCI and 90 minutes after PCI
Effectiveness of the method used in regards to development of heart failure. | During in hospital stay up to 36 hours
  Development of acute heart failure after PCI during hospital admission.
Effectiveness of the method used in regards to mortality. | During in hospital stay up to 36 hours
  Death during hospital stay post-PCI.
Safety of the method used in regards to bleeding. | During in hospital stay up to 36 hours
  Bleeding events will be noted and classified according to BARC (Bleeding Academic Research Consortium) bleeding score during hospital stay post-PCI
Safety of the method used in regard to development of arrhythmia. | During in hospital stay up to 36 hours
  Development of arrhythmia post-PCI will be noted and the type of arrhythmia will be identified.

SECONDARY OUTCOMES:
Follow up post-PCI by trans-thoracic Echo | During in hospital stay up to 36 hours
  To estimate the ejection fraction on discharge.
Follow up post-PCI in regards to MACE (Major adverse cardiac events) | 3 and 6 months after procedure
  The development of MACE: Death, myocardial infarction, hospitalization due to heart failure, recurrent PCI or CABG.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abdelghany, Prof, Study Director — Assiut University; Ayman Khairy, Prof, Study Director — Assiut University

REFERENCES:
- [Background] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Background] Miranda-Guardiola F, Rossi A, Serra A, Garcia B, Rumoroso JR, Iniguez A, Vaquerizo B, Triano JL, Sierra G, Bruguera J; Spanish AMIcath Registry. Angiographic quantification of thrombus in ST-elevation acute myocardial infarction presenting with an occluded infarct-related artery and its relationship with results of percutaneous intervention. J Interv Cardiol. 2009 Jun;22(3):207-15. doi: 10.1111/j.1540-8183.2009.00464.x. Epub 2009 Apr 14. PMID 19490354
- [Background] Kumar V, Sharma AK, Kumar T, Nath RK. Large intracoronary thrombus and its management during primary PCI. Indian Heart J. 2020 Nov-Dec;72(6):508-516. doi: 10.1016/j.ihj.2020.11.009. Epub 2020 Nov 19. PMID 33357638
- [Background] Yip HK, Chen MC, Chang HW, Hang CL, Hsieh YK, Fang CY, Wu CJ. Angiographic morphologic features of infarct-related arteries and timely reperfusion in acute myocardial infarction: predictors of slow-flow and no-reflow phenomenon. Chest. 2002 Oct;122(4):1322-32. doi: 10.1378/chest.122.4.1322. PMID 12377860
- [Background] Pradhan A, Bhandari M, Vishwakarma P, Sethi R. Deferred Stenting for Heavy Thrombus Burden During Percutaneous Coronary Intervention for ST-Elevation MI. Eur Cardiol. 2021 Mar 30;16:e08. doi: 10.15420/ecr.2020.31. eCollection 2021 Feb. PMID 33897834
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Chesebro JH, Knatterud G, Roberts R, Borer J, Cohen LS, Dalen J, Dodge HT, Francis CK, Hillis D, Ludbrook P, et al. Thrombolysis in Myocardial Infarction (TIMI) Trial, Phase I: A comparison between intravenous tissue plasminogen activator and intravenous streptokinase. Clinical findings through hospital discharge. Circulation. 1987 Jul;76(1):142-54. doi: 10.1161/01.cir.76.1.142. PMID 3109764
- [Background] Vranckx P, White HD, Huang Z, Mahaffey KW, Armstrong PW, Van de Werf F, Moliterno DJ, Wallentin L, Held C, Aylward PE, Cornel JH, Bode C, Huber K, Nicolau JC, Ruzyllo W, Harrington RA, Tricoci P. Validation of BARC Bleeding Criteria in Patients With Acute Coronary Syndromes: The TRACER Trial. J Am Coll Cardiol. 2016 May 10;67(18):2135-2144. doi: 10.1016/j.jacc.2016.02.056. PMID 27151345